CLINICAL TRIAL: NCT06283459
Title: Phase 1/2, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of a DNA Vaccine, IMNN-101, Administered as a Single Dose in Healthy Adults Previously Vaccinated Against SARS-CoV-2
Brief Title: Study to Evaluate the Safety & Immunogenicity of IMNN-101 Administered in Healthy Adults Previously Vaccinated Against SARS-CoV-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imunon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 301-23-101
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMNN-101 (Experimental): Participants will receive a single intramuscular (IM) dose of IMNN-101 on Day 0 in the deltoid muscle.
  IMNN-101 is for intramuscular injection only.
  Interventions: Biological: IMNN-101

INTERVENTIONS:
Biological: IMNN-101 — IMNN-101 is a DNA vaccine encoding SARS-CoV-2 Omicron XBB.1.5 spike antigen. The drug product is a suspension of the DNA plasmid formulated with the facilitating agent, bis-(aza-18-crown-6)-poloxamer (Crown poloxamer, CP), and adjuvant AlPO4.

SUMMARY:
This is an open-label phase 1/2, dose-escalation study. Participants will receive a single intramuscular (IM) dose of IMNN-101 on Day 0 in the deltoid muscle and will be followed through 12 months post-vaccination (through Study Day 365).

DETAILED DESCRIPTION:
This is an open-label phase 1/2, dose-escalation study. Participants will receive a single intramuscular (IM) dose of IMNN-101 on Day 0 in the deltoid muscle and will be followed through 12 months post-vaccination (through Study Day 365).

Phase 1: A total of twenty-four (24) participants will be enrolled into one of three groups listed below:

Group 1 (8 participants) - 0.25 mL at 2 mg/ml of IMNN-101 DNA to be administered as 0.5 mg dose intramuscularly (IM) at Day 0

Group 2 (8 participants) - 0.50 mL at 2 mg/ml of IMNN-101 DNA to be administered as 1.0 mg dose intramuscularly (IM) at Day 0

Group 3 (8 participants) - 1.0 mL at 2 mg/ml of IMNN-101 DNA to be administered as 2.0 mg dose intramuscularly (IM) at Day 0

To assess early safety signals for this Phase 1 study, vaccination will proceed in a staged fashion. Sentinel participant dosing will begin with 4 participants in Group 1 (0.25 mL). If no halting rules have been met after Group 1 sentinels complete Day 7, then the remaining 4 participants in Group 1 may enroll and sentinel dosing will begin with 4 participants in Group 2 (0.5 mL). If no halting rules have been met after Group 2 sentinels complete Day 7, then the remaining 4 participants in Group 2 may enroll and sentinel dosing will begin with 4 participants in Group 3 (1.0 mL). If no halting rules have been met after Group 3 sentinels complete Day 7, then the remaining 4 participants in Group 3 may enroll.

Phase 2: Once a review of the safety and immunogenicity is completed in Phase 1 then an expansion Phase 2 will commence utilizing the recommended Phase 2 dose (RP2D). Fifty (50) healthy participants meeting eligibility criteria will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to complete the informed consent process, including an Assessment of Understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered correctly.
2. 18-65 years old, inclusive, on day of enrollment.
3. Agrees to comply with planned study procedures and be available for clinic follow-up through the last clinic visit.
4. Willing to disclose prior SARS-CoV-2 infection and/or prior vaccination (via COVID-19 vaccination card or other reliable record).
5. Previously received at least one COVID-19 immunization with the last dose > 4 months prior to enrollment.
6. Willing to forego any non-study vaccinations from time of study enrollment to at least 28 days from the dose of study vaccination.
7. Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the 302-23-101 study team are required.
8. In good general health according to the clinical judgement of the site investigator.
9. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator. Clinically significant hematology and/or blood chemistry laboratory results that meet the definition of Grade ≥2 abnormality will prevent the inclusion in the trial. Investigators should reference Appendix D, FDA guidance, Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
10. Body mass index of 18-35 kg/m2, inclusive, at screening
11. Negative results for HIV infection by an (US) Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
12. Negative for anti-Hepatitis C antibodies (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV antibodies are detected.
13. Negative for Hepatitis B surface antigen.
14. For a volunteer assigned female sex at birth and capable of becoming pregnant or a volume assigned male sex at birth:

Volunteers who were assigned female sex at birth and are of reproductive potential must agree to use an acceptable method of contraception from at least 21 days prior to study Day 0 until at least 90 days after vaccination. Volunteers who are physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with individuals born male must use an acceptable method of contraception during this period. Acceptable methods of contraception include a sterile sexual partner, hormonal contraceptives (combined estrogen and progestogen containing), hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, sexual abstinence.

Has negative β-HCG (beta human chorionic gonadotropin) pregnancy test (urine or serum) at screening and prior to study product administration.

Sexually active participants assigned male sex at birth must be willing to use an effective method of contraception (i.e., condoms or be anatomically sterile) from Day of Injection through Day 28.

Exclusion Criteria:

1. Positive RT-PCR test for SARS-CoV-2 within two days of screening.
2. Known history of SARS-CoV-2 infection within 3 months of screening.
3. COVID-19 monoclonal antibody-based treatment within 3 months of screening.
4. Is currently participating in another COVID-19 vaccine study and is in the 12-month follow up period for that vaccine or has participated in a study with an investigational product within 30 days preceding Day 0.
5. Fever (tympanic temperature > 37.5°C), dry cough, fatigue, nasal obstruction, runny nose, sore throat, myalgia, diarrhea, shortness of breath or dyspnea within 14 days prior to vaccine administration.
6. Volunteers with abnormal indicators at screening, such as blood biochemistry, blood routine and urine routine deemed to be clinically significant by the investigator.
7. Volunteers with a history of myocarditis or pericarditis and/or a history of cardiac insufficiencies class III and IV of the New York Heart Association (NYHA) Classification.
8. History of severe allergic reactions (such as acute anaphylaxis, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain) or allergy to any pertinent components of IMNN-101.
9. History of significant CNS disease such as prior convulsions, epilepsy, encephalopathy, or a history of severe mental illness.
10. Diagnosed with severe liver and/or kidney diseases, uncontrollable hypertension, diabetic complications, malignant tumors, acute viral or bacterial infections or acute onset of any chronic disease.
11. Diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia, or other autoimmune diseases.
12. History of coagulation dysfunction (e.g., coagulation factor deficiency, coagulation disease).
13. Received any vaccine within 28 days prior to the study vaccine.
14. Receiving immunotherapy or inhibitor therapy within 3 months (consistently oral or infusion for more than 14 days).
15. Received systemic immunosuppressants within 4 months prior to vaccination or anticipating the need for immunosuppressant at any time during participation in the study. Topical or inhaled treatment is allowed if not used within 14 days prior to vaccination.
16. Received any blood products within 3 months before IMNN-101 administration.
17. History of alcohol or drug abuse within 3 years before first vaccination.
18. Has donated >450 mL of whole blood within 28 days prior to vaccination.
19. History of anaphylaxis or angioedema, including but not limited to a history of anaphylaxis after receipt of any vaccine.
20. Any condition that, in the opinion of the investigator, would (a) pose a health risk to the volunteer if enrolled or (b) could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
21. Volunteer who is breast-feeding or pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with local and systemic reactogenicity adverse events and all adverse events | 1 month
  Local and systemic reactogenicity signs and symptoms for a minimum of seven days following receipt of study product. Laboratory measures of safety. All adverse events (AEs) for thirty days after receipt of study vaccination.
  All serious adverse events (SAEs), medically attended adverse events (MAAEs), adverse events of special interest (AESIs), and AEs leading to early participant withdrawal or permanent discontinuation will be collected throughout the study.
Number of participants with geometric mean titer (GMT) of the serum neutralizing antibody (Nab) against the Omicron XBB.1.5 strain. | 12 months
  Geometric mean titer (GMT) of the serum neutralizing antibody (Nab) against the Omicron XBB.1.5 strain at baseline and at 0.5, 1 month, 3 months, 6 months, 9 months, and 12 months.

SECONDARY OUTCOMES:
Number of participants with GMT of serum spike binding IgG antibodies | 12 months
  GMT of serum spike binding IgG antibodies at baseline and at 0.5, 1 month, 3 months, 6 months, 9 months, and 12 months.
Number of participants with a magnitude and phenotype of cytokine producing S protein-specific T cells, as measured by flow cytometry and/or ELISpot. | 9 months
  Magnitude and phenotype of cytokine producing S protein-specific T cells, as measured by flow cytometry and/or ELISpot at baseline and at 1 month, 3 months, 9 months (Phase-1) and at baseline and at 1 month, 9 months (Phase-2).
Number of participants with seroresponse rate (SRR). | 28 days
  Seroresponse rate (SRR), defined as a ≥ 4-fold increase of Nab or binding antibody titers 28 days after vaccine administration (relative to pre-vaccination baseline). The geometric mean fold rise (GMFR) in IgG titers of 28 days after vaccine administration, relative to baseline, for both Nab and binding antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Faller, MD, Study Director — Imunon
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - DM Clinical Research, Philadelphia, Pennsylvania